CLINICAL TRIAL: NCT03570450
Title: Regenerative Stem Cell Therapy for Stroke in Europe 1
Brief Title: Regenerative Stem Cell Therapy for Stroke in Europe 1-RESSTORE1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Horizon 2020 - European Commission (Other); University Grenoble Alps (Other); Servicio Madrileño de Salud, Madrid, Spain (Other); St. Anne's University Hospital Brno, Czech Republic (Other); Andaluz Health Service (Other Government); University of Glasgow (Other); University of Eastern Finland (Other); Etablissement Français du Sang (Other); Tampere University (Other); Histocell SL, Spain (Unknown); Oy Medfiles Ltd (Industry); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Hospices Civils de Lyon (Other); Association Groupe ESSEC (Other); NOVADISCOVERY SAS, France (Unknown); Finovatis (Other); Centre Hospitalier Universitaire de Besancon (Other); Assistance Publique - Hôpitaux de Paris (Other); University Hospital, Toulouse (Other); University Hospital, Bordeaux (Other); University Hospital, Caen (Other); Fundación Instituto de Estudios de Ciencias de la Salud de Castilla y León (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Servicio de Salud de Castilla La Mancha, Albacete, Spain (Unknown); Servicio Gallego de Salud (Other Government); Pirkanmaa Hospital District, Tampere, Finland (Unknown); Hospital Vall d'Hebron (Other); Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other); CH Sainte-Anne, Paris, France (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 38RC17.312
Record Dates: First submitted 2018-04-18; First posted 2018-06-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Stroke
Keywords: Cell therapy; stem cell; transplantation; graft; recovery; repair; stroke; msesenchymal stem cell; regenerative
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: * Dose escalation from 1.10^6 cells/kg to 3.10^6 cells/kg (phase 1a, non randomized, open-label);
  * Effect-dose: 3.10^6 cells/kg + placebo (phase 1b, randomized, double blind);
  Phase Ia: n = 15 patients; Phase Ib: n = 80 patients
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Adipose derived Stem Cells - 1.10^6cells/kg (Experimental): ADSC, single, IV, 1.10^6cells/kg
  Interventions: Drug: Adipose derived Stem Cell
- Adipose derived Stem Cells - 2.10^6cells/kg (Experimental): ADSC, single, IV, 2.10^6cells/kg
  Interventions: Drug: Adipose derived Stem Cell
- Adipose derived Stem Cells - 2,5.10^6cells/kg (Experimental): ADSC, single, IV, 2,5.10^6cells/kg
  Interventions: Drug: Adipose derived Stem Cell
- Adipose derived Stem Cells - 3.10^6cells/kg (Experimental): ADSC, single, IV, 3.10^6cells/kg
  Interventions: Drug: Adipose derived Stem Cell
- placebo (Placebo Comparator): Placebo
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Adipose derived Stem Cell — 4 doses
  Other Names: ADSC
  Arms: Adipose derived Stem Cells - 1.10^6cells/kg; Adipose derived Stem Cells - 2,5.10^6cells/kg; Adipose derived Stem Cells - 2.10^6cells/kg; Adipose derived Stem Cells - 3.10^6cells/kg
Other: placebo — placebo
  Arms: placebo

SUMMARY:
Stroke is the second leading cause of death in the world population. When not fatal, stroke often results in disability, and secondary health problems affecting not only patients but also their families. Building on emerging preclinical and pilot clinical evidences, RESSTORE will focus on the clinical assessment of regenerative cell therapy to improve stroke recovery and patients quality of life.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria are similar in the phase 1a (RESSTORE 1a, Toxicity study) and in the phase 1b (RESSTORE 1b, Dose-effect study).

* Male or female > 18-year-old
* Hemispheric ischemic stroke (> 1.5 cm on 2 imaging slices) (i.e. non "lacunar" stroke) Admitted to the stroke unit within the first 24h after stroke onset
* Patient must be included within 1st and 2nd day after stroke onset (signature of informed consent and randomization) (i.e. between 24 hours and 48 hours from stroke onset) and must be able to receive investigation treatment within the first week.
* NIHSS > or equal to 7 including motor score (upper, lower limbs and hand) > or equal to 3
* No decompressive craniectomy procedure planned or performed
* Patient able to follow a rehabilitation program
* Modified Rankin scale = 0 before stroke onset
* Obtained signed informed consent from patient or legally acceptable representative
* Negative pregnancy test for women of child-bearing age.

Non Inclusion Criteria:

Non-inclusion criteria are similar in the phase 1a (RESSTORE 1a, Toxicity study) and the phase 1b (RESSTORE 1b, Dose-effect study).

* Contraindication for MRI
* Coma (score of 2 or more on item 1a of the NIHSS related to awareness)
* Evidence on neuroimaging (CT or MRI) of a brain tumour, cerebral oedema with midline shift and a clinically significant compression of ventricles, cerebellar or brainstem infarction, or subarachnoid haemorrhage, or intracerebral parenchymal hematoma (petechial small haemorrhages are NOT a non-inclusion criteria)
* Severe leucoariosis
* Previous stroke
* Active endocarditis, pneumonia, AIDS, active hepatic disease due to HBV or HCV (a controlled infection is NOT a non-inclusion criteria)
* Active inflammatory and/or auto-immune diseases (such as Crohn disease, lupus, rheumatoid polyarthritis, renal or liver immune pathology)
* History of cancer
* Pre-existing dementia
* A health status, any clinical condition (eg, short life expectancy, and coexisting disease) or other characteristic that precludes appropriate diagnosis, treatment, or follow-up in the trial
* Surgical or endovascular procedure planned in the following 3 months
* Pregnancy / Breast feeding (women of childbearing age should have a negative pregnancy test prior to inclusion)
* Patients who are participating in another therapeutic trial or who have previously participated in a biotherapy trial
* Non-membership to a social security scheme
* Inability or unwillingness of the individual or their legal guardian/representa tive to provide written informed consent, according to national regulations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2018-06-02 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Phase Ia (Toxicity study) | 7 days after stroke onset
  cell-related serious adverse event
Phase Ib (Dose-effect study) | 6 months after stroke onset
  modelling the dose-effect

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability | through study completion (2 years)
  Adverse events report and mortality over 2 years
Functionnal recovery | through study completion (2 years)
  NIHSS Evolution (0-42) over 2 years
Post stroke handicap | through study completion (2 years)
  Modified Rankin scale (0-6) over 2 years
Motor recovery | over 6 months post-stroke
  Fugl Meyer score (0-226) assessed by physiotherapist over 6 months post-stroke
fMRI recovery | at 6 months post-stroke
  activation fMRI and resting state fMRI at 6 months after stroke
Blood biomarkers for stroke recovery | at 6 months post-stroke
  selection of candidate biomarkers for stroke recovery

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Detante, MD PhD, Principal Investigator — University Hospital Grenoble-Alpes
Locations (1):
- CHU Grenoble Aples, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Legris L, Moisan A, Jaillard A, Bonnet L, Moulin T, Sibon I, Touze E, Favre-Wiki I, Cordonnier C, Dellaschiava L, Mazighi M, Rosso C, Alamowitch S, Calvet D, Barbieux-Guillot M, Roux S, Mojallal AA, Boucher F, Thuriot A, Soulard J, Naegele B, Perennou D, Roustit M, Putkaradze Z, Hommel M, Lehmann A, Colombat J, Chorfa F, Maucort-Boulch D, Lamalle L, Grand S, Krainik A, Detante O. Regenerative stem cell therapy for stroke in Europe (RESSTORE): a multicenter randomized controlled efficacy clinical trial. Front Stroke. 2024 Sep 27;3:1416490. doi: 10.3389/fstro.2024.1416490. eCollection 2024. PMID 41542240